CLINICAL TRIAL: NCT02052089
Title: Prospective Randomized Clinical and Radiologic Study for the Treatment of Lateral Epicondylosis; Comparison Among PRP (Platelet-Rich Plasma) , Prolotherapy, Physiotherapy and ESWT (Extracorporeal Shockwave Therapy)
Brief Title: Comparative Study for the Optimal Treatment Method of Lateral Epicondylosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: CM Chungmu Hospital (Other)
Responsible Party: Principal Investigator, Sang-Hoon Lhee, Director of CM Chungmu Hospital, CM Chungmu Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CMH-2014-04
Record Dates: First submitted 2014-01-22; First posted 2014-01-31 (Estimated); Last update posted 2014-01-31 (Estimated); Status verified 2014-01

CONDITIONS: Tennis Elbow
Keywords: Tennis Elbow; lateral epicondylosis; lateral epicondylitis; Platelet-Rich Plasma; Extracorporeal Shockwave Therapy; Prolotherapy; Physiotherapy
MeSH Terms: conditions — Tennis Elbow | interventions — Physical Therapy Modalities; Rehabilitation; Extracorporeal Shockwave Therapy; Prolotherapy

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Physiotherapy (Active Comparator): patients were educated to do stretching and eccentric strengthening exercise of wrist extensor muscles
  Interventions: Procedure: physiotherapy
- extracorporeal shockwave therapy (Experimental): patients were treated with 3 sessions of high-energy shock wave therapy ESWT (Evotron, Switech medical, Kreuzlingen, CH) in 2 weeks interval. Total energy flux density ranged from 0.1 to 0.14 mJ/mm2 (1500 impulses). Shockwave was targeted over lateral epicondyle where maximum tenderness was located.
  Interventions: Procedure: extracorporeal shockwave therapy
- Prolotherapy (Experimental): injection of 20% dextrose (3cc mixed with 0.3cc of lidocaine) to ECRB tendon was done under ultrasound guidance
  Interventions: Procedure: prolotherapy
- Platelet-rich plasma (Experimental): 3 cc of PRP (Harvest SmartPReP 2 APC 30 Process Kit, Harvest Technologies, Plymouth, MA) was injected into ECRB tendon under ultrasound guidance
  Interventions: Procedure: platelet-rich plasma

INTERVENTIONS:
Procedure: physiotherapy — Physiotherapy is the treatment of a wide range of conditions and injuries to the body through the use of various forms of passive mobilisation, massage, electrotherapy and exercises.
  Other Names: Physical Therapy; Rehabilitation
  Arms: Physiotherapy
Procedure: extracorporeal shockwave therapy — Extracorporeal shockwave therapy (ESWT) is noninvasive procedure, and has been shown to be effective in the treatment of chronic tendon pathology in the elbow, shoulder and plantar fascia. Shock wave therapy is traditionally categorized as either low energy (<0.2 mJ/mm2) or high energy (>0.2 mJ/mm2). Rompe, et al have hypothesized that there is an overstimulation of nerve fibers, resulting in an immediate analgesic effect (hyperstimulation analgesia). Physical effects on cell permeability and induction of diffusible radicals have also been postulated to cause disruption of the tendon tissue, resulting in induction of a healing process.
  Other Names: ESWT
  Arms: extracorporeal shockwave therapy
Procedure: prolotherapy — Prolotherapy has been defined as the iatrogenic stimulation of wound healing and tissue repair through the injection of an irritant solution into damaged ligaments and tendons. Prolotherapy solutions are purported to initiate an inflammatory cascade at the site of injection, which induces fibroblast proliferation and subsequent collagen synthesis, resulting in a tighter and stronger ligament or tendon. The primary mechanism of action of prolotherapy is to induce a small inflammatory response to promote adequate healing or more viable scar tissue formation that results in stronger fibrous tissue at the lateral epicondyle, which leads to improved function and reduced pain.
  Arms: Prolotherapy
Procedure: platelet-rich plasma — Platelet-rich plasma (PRP) is defined as an autologous concentration of human platelets in a small volume of plasma which is mechanically treated to increase the concentration of platelets compared to whole blood. The supraphysiological concentration of platelets will provide a locally increased concentration of growth factors and cytokines that are contained within the platelets themselves.Based on these concepts, it is believed that PRP can augment or stimulate healing with the same biologic healing process that normally occurs in the human body after injury.
  Other Names: PRP
  Arms: Platelet-rich plasma

SUMMARY:
The purpose of this study is to find the optimal treatment method for chronic lateral epicondylosis, and focused on the 'healing mechanism' and 'pain modulation' of degenerated tendon.The hypothesis is that there will be significant difference between treatment groups and control group (physiotherapy) and also there will be significant difference among treatment groups.

DETAILED DESCRIPTION:
231 patients were randomized using a Random Sequence Generator (Random.org) into 4 groups: Group A (physiotherapy as a control, n=58), Group B (ESWT, n=62), Group C (Prolotherapy, n=56) and Group D (PRP, n=55). In group A, patients were educated to do stretching and eccentric strengthening exercise of wrist extensor muscles. In group B patients were treated with 3 sessions of high-energy shock wave therapy ESWT (Evotron, Switech medical, Kreuzlingen, CH) in 2 weeks interval. Total energy flux density ranged from 0.1 to 0.14 mJ/mm2 (1500 impulses). Shockwave was targeted over lateral epicondyle where maximum tenderness was located. In group C, injection of 20% dextrose (3cc mixed with 0.3cc of lidocaine) to ECRB tendon was done under ultrasound guidance and in group D, 3 cc of PRP (Harvest SmartPReP 2 APC 30 Process Kit, Harvest Technologies, Plymouth, MA) was injected into ECRB tendon under ultrasound guidance. 22G needle was used for injection in group C and D. The primary outcome measure is DASH scoring system which is recorded on the initial, 3rd, 6th, 18th and 24th month. Secondary outcome measures were ultrasonography (measured on initial, 6th and 24th month) and SSS (Subjective Satisfaction Score) measured on initial and 24th month. After 24 months from the last procedure, all serial questionnaires and physician-filled-SSS sheets were gathered and analyzed by a one-way analysis of variance and Scheffe post-test. A value of p<0.01 was considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* 35 to 80 years of age
* history of elbow pain in the region of the lateral epicondyle for more than 6 months
* more than 3 months of treatment for lateral epicondylosis before enrollment in the study with no subjective improvement
* pain on resisted extension of wrist
* local tenderness to palpation at the lateral epicondyle
* confirmed as lateral epicondylosis on ultrasound imaging

Exclusion Criteria:

* history of steroid or botulinum injection(s) within 6 months before study enrollment
* other elbow pathology including nerve compression, previous elbow fracture, limited elbow range of motion, abnormal simple radiographic findings, history of elbow surgery and inflammatory arthropathies
* upper extremity pain or discomforts from shoulder or wrist or hand

Ages: 35 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 231 (Actual)
Dates: Start 2009-03; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
DASH scoring system to measure the changes in the upper extremity function | upon initial examination, 3-month follow-up, 6-month follow-up, 18-month follow-up, 24-month follow-up
  The DASH is intended to measure how much difficulty a subject has when performing common functional tasks and activities. The DASH consists of a 30-item questionnaire with 5 response options for each item with a scale ranging from 0, which indicates "least disability," to 100, which indicates "most disability." It incorporates questions related to functional limitations, symptoms, and psychosocial problems. The DASH has been well validated and has a smaller standard error of measurement and a validity comparable to that of joint-specific measures. Based on our preliminary study, grand mean of DASH score was set to 26.05, and we decided that 8 points difference of DASH score will be the minimum detectable change.

SECONDARY OUTCOMES:
SSS (Subjective Satisfaction Score) | upon initial examination and on the 24th month
  SSS (Subjective Satisfaction Score) which is answered by following question.
  " How do you feel now compared to the condition before treatment in terms of satisfaction"
  0 - It is worse. Not satisfied at all
  1. - There are no change and still it is as uncomfortable as before. Not satisfied at all
  2. - Slightly improved but less than 50% of the pain is subsided. Not so satisfied.
  3. - About 50% of the pain or discomfort is gone. Slightly satisfied, but not so much
  4. - About 75% of the pain or discomfort is gone. Definitely better. Satisfied.
  5. - More than 75% of the pain or discomfort is gone. Much better and very satisfied.
ultrasonography to asses changes in tendon pathology | upon initial examination, 6th month and 24th month
  In our study, we measure the changes in the hypoechogenicity of the tendon and via color doppler to determine the amount of vascularity noted in the tendon.Ultrasonography (US) is an important tool in sports medicine and rheumatology, and a common outcome measure in clinical trials. In general, US is a noninvasive, widely available, and inexpensive imaging technique for assessing tendon pathology. The high acoustic contrast with the surrounding tissue makes tendons particularly suitable for ultrasonographic examination. US findings in tendinopathy in general are characterized by increased tendon size, Doppler activity, irregularity of the fibrillar appearance, focal hypoechoic areas, and calcifications.

CONTACTS AND LOCATIONS:
Overall Officials: Sang-Hoon Lhee, MD PhD, Principal Investigator — CM Chungmu Hospital
Locations (1):
- CM Chungmu Hospital, Seoul, Yeongdeungpo-gu, South Korea

REFERENCES:
- [Derived] Karjalainen TV, Silagy M, O'Bryan E, Johnston RV, Cyril S, Buchbinder R. Autologous blood and platelet-rich plasma injection therapy for lateral elbow pain. Cochrane Database Syst Rev. 2021 Sep 30;9(9):CD010951. doi: 10.1002/14651858.CD010951.pub2. PMID 34590307